CLINICAL TRIAL: NCT04249531
Title: Pharmacokinetic Evaluation and Local Tolerability of Dry Powder Amikacin Via the Cyclops™ in Patients With Drug Susceptible Tuberculosis
Brief Title: Pharmacokinetic Evaluation and Local Tolerability of Dry Powder Amikacin Via the Cyclops™
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Onno Akkerman, Principal investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Amika-01
Record Dates: First submitted 2019-08-19; First posted 2020-01-31 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amikacin (Experimental): Patients will receive once amikacin i.v. 7,5 mg/kg in the first week
  Interventions: Drug: Amikacin Inhalation Dry Powder; Drug: Amikacin Injectable Product

INTERVENTIONS:
Drug: Amikacin Inhalation Dry Powder — Patient will inhale the weeks after iv amikacin, dry powder amikacin per inhalation once 400 mg, next week once 700 mg and the last week 1000 mg
Drug: Amikacin Injectable Product — patient wil receive one dose of 400 mg amikacine intravenously in week 1

SUMMARY:
Rationale: Multidrug-resistant tuberculosis (MDR-TB) is defined as tuberculosis resistant to isoniazid and rifampicin. The incidence of MDR-TB worldwide is 3.9% for new cases and 21% for previously treated cases. However, the incidence of previously treated cases can rise to above 50% in eastern European countries. With increasing frequency of MDR-TB (and even extensively drug-resistant types), morbidity and mortality due to TB fail to decline worldwide. Amikacin, one of the drugs against MDR-TB, has the most potent effect when reaching a high peak serum concentration and this means that high doses have to be administered. Treatment with amikacin by inhalation would be a tremendous advantage due to the high local dose in the lungs, obtaining high local levels without the possible toxicity due to high serum levels. With the currently available inhalation techniques these local levels cannot be reached easily.

In this protocol, the investigators will perform a pharmacokinetic and local tolerability study of dry powder amikacin using the Cyclops™ in patients with drug susceptible tuberculosis.

Objective:

* primary objective is to investigate the pharmacokinetic properties of dry powder amikacin at different dosages and compare the peak serum values to a single i.v. dose.
* secondary objective is to assess the local tolerability of dry powder amikacin via the Cyclops™ at different dosages.

Study design: single center, active control, ascending dose response study Study population: 8 patients with DSTB. Main study parameters/endpoints: the following pharmacokinetic parameters: actual dose (dose minus remainder in inhaler after inhalation), AUC0-24 (area under the curve from 0-24 h), Cmax (maximum serum concentration), Tmax (time to maximum serum concentration).

For the local tolerability the following procedures will be done, drop of FEV1 of >15 % (lung function measurement) and any other reported adverse event are all considered critical to decide on proceeding into a phase 2B (and/or a phase 3) trial.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participants included in this study are patients with DSTB, who are admitted at the Tuberculosis Center Beatrixoord. They will receive 3 different doses of amikacin using the DPI with (at least) one week in between doses, they will also receive one dose of intravenous amikacin. Before using the dry powder inhaler (DPI) they will receive instructions and their inspiratory flow will be tested. Before each test dose an indwelling cannula will be inserted and before and after each test dose in total 9 blood samples will be collected. To investigate local tolerability, lung function tests will be performed and the occurrence of adverse events will be scored.

DETAILED DESCRIPTION:
Rationale: Multidrug-resistant tuberculosis (MDR-TB) is defined as tuberculosis resistant to isoniazid and rifampicin. The incidence of MDR-TB worldwide is 3.9% for new cases and 21% for previously treated cases. However, the incidence of previously treated cases can rise to above 50% in eastern European countries. With increasing frequency of MDR-TB (and even extensively drug-resistant types), morbidity and mortality due to TB fail to decline worldwide. Cornerstones of MDR-TB treatment are aminoglycosides, like amikacin, and fluoroquinolones. Amikacin is given intravenously for 6-8 months in the usual MDR-TB treatment. Since 2016 it can also be given for 4-6 months in the short-course treatment for MDR-TB. In many countries, this implicates long hospital admissions for the patients, as well as problems in venous access, often necessitating surgical insertion of venous access ports. Amikacin has the most potent effect when reaching a high peak serum concentration and this means that high doses have to be administered. Treatment with amikacin by inhalation would be a tremendous advantage due to the high local dose in the lungs, obtaining high local levels without the possible toxicity due to high serum levels. With the currently available inhalation techniques these local levels cannot be reached easily.

In this protocol, the investigators will perform a pharmacokinetic and local tolerability study of dry powder amikacin using the Cyclops™ in patients with drug susceptible tuberculosis (DSTB, as opposed to MDRTB).

Objective:

* primary objective is to investigate the pharmacokinetic properties of dry powder amikacin at different dosages and compare the peak serum values to a single i.v. dose.
* secondary objective is to assess the local tolerability of dry powder amikacin via the Cyclops™ at different dosages.

Study design: single center, active control, ascending dose response study Study population: 8 patients with DSTB. Main study parameters/endpoints: The following pharmacokinetic parameters will be calculated: actual dose (dose minus remainder in inhaler after inhalation), AUC0-24 (area under the curve from 0-24 h), Cmax (maximum serum concentration), Tmax (time to maximum serum concentration).

For the local tolerability of the inhalation of dry powder amikacin the following procedures will be done, drop of FEV1 of >15 % (lung function measurement) and any other reported adverse event are all considered critical to decide on proceeding into a phase 2B (and/or a phase 3) trial.

The inspiratory parameters during the inhalation maneuver are critical to explore predictors for drug exposure. The following parameters will be calculated: dPmax (maximum pressure drop), Vi (inhaled volume), Ti (total inhalation time), PIF (peak inspiratory flow rate), MIF (mean inspiratory flow rate) and the FIR (average flow increase rate between 20% and 80% of PIF) Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participants included in this study are patients with DSTB, who are admitted at the Tuberculosis Center Beatrixoord. They will receive 3 different doses of amikacin using the DPI with (at least) one week in between doses, they will also receive one dose of intravenous amikacin. Before using the dry powder inhaler (DPI) they will receive instructions and their inspiratory flow will be tested. Before each test dose an indwelling cannula will be inserted and before and after each test dose in total 9 blood samples will be collected. To investigate local tolerability, lung function tests will be performed and the occurrence of adverse events will be scored.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosed with DSTB, either by culture or molecular testing
* Obtained written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Subjects with known or suspected (by spontaneous reporting or by active questioning) renal, auditory, vestibular or neuromuscular dysfunction.
* History of adverse events on previous amikacin or other aminoglycoside use (by spontaneous reporting nor by active questioning)
* Concurrent use of cyclosporin, cisplatin, amfotericin B, cephalosporins, polymyxins and vancomycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The actual dose will be calculated | 1 day
  actual dose
The AUC0-24 will be calculated | 1 day
  AUC0-24
The Cmax will be calculated | 1 day
  Cmax
The Tmax will be calculated | 1 day
  Tmax
Local tolerability of the inhalation of dry powder amikacin will be established. | 1 day
  drop of forced expiratory volume in 1 second (FEV1)FEV1 of >15 % (lung function measurement)
The tolerability of the inhalation of dry powder amikacin will be established | 1 day
  questioning and registration of adverse events.

SECONDARY OUTCOMES:
The dPmax (maximum pressure drop) will be measured | 15 - 30 minutes
  dPmax
The Vi (inhaled volume) will be measured | 15 - 30 minutes
  Vi (inhaled volume)
The Ti (total inhalation time) will be measured | 15 - 30 minutes
  Ti (total inhalation time)
The PIF (peak inspiratory flow rate) will be measured | 15 - 30 minutes
  PIF (peak inspiratory flow rate)
The MIF (mean inspiratory flow rate) will be measured | 15 - 30 minutes
  MIF (mean inspiratory flow rate)
The FIR (average flow increase rate between 20% and 80% of PIF) will be measured | 15 - 30 minutes
  FIR (average flow increase rate between 20% and 80% of PIF)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands